CLINICAL TRIAL: NCT03474900
Title: Elastic Stable Intramedullary Nailing of Forearm Shaft Fractures by Titanium Compared With Biodegradable Nails: Results of a Prospective Randomized Trial in Children With at Least Two Years of Follow-up
Brief Title: Biodegradable Versus Titanium Nailing in Forearm Shaft Fractures in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaakko Sinikumpu (Other)
Collaborators: Oulu University Hospital (Other); Bioretec Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Jaakko Sinikumpu, Head of childhood fracture and sport injury study, M.D., Ph.D., Oulu University Hospital
Organization: Oulu University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Oulu University Hospital
Record Dates: First submitted 2018-01-05; First posted 2018-03-23 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Forearm Fracture
Keywords: intramedullary nailing; randomised controlled trial; biodegradable; children; forearm shaft fractures

STUDY DESIGN:
Intervention Model Description: The patients were randomised to 2 groups, titanium nailing or biodegradable nailing.
Masking Description: The patient was informed about the treatment method that he or she was randomised. The operating surgeon knew the group and treatment that the patient belonged to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLGA implant, Bioretec ltd. Finland (Experimental): Treatment with biodegradable elastic stable intramedullary nail in unstable forearm shaft fracture in paediatric population
  Interventions: Device: PLGA implant, Bioretec ltd. Finland
- Titanium elastic stable nail (Active Comparator): Treatment with titanium elastic stable intramedullary nail in unstable forearm shaft fracture in paediatric population
  Interventions: Device: Titanium elastic stable nail

INTERVENTIONS:
Device: PLGA implant, Bioretec ltd. Finland — The investigational implant is an ultra-high-strength biodegradable intramedullary (IM) nail of poly(lactide-co-glycolide) (PLGA)/tricalcium-phosphate (β-TCP) which was manufactured by Bioretec Ltd. (Hartmaninkatu 2, Tampere, Finland)
  Other Names: Biodegradable elastic stable intramedullary nail
  Arms: PLGA implant, Bioretec ltd. Finland
Device: Titanium elastic stable nail — Elastic stable intramedullary nail to stabilize unstable forearm shaft fractures in children
  Other Names: elastic stable intramedullary nail
  Arms: Titanium elastic stable nail

SUMMARY:
There are disadvantages in Elastic Stable Intramedullary Nailing (ESIN) of forearm shaft fractures, such as soft tissue irritation and the need of implant removal. A new mini-invasive technique of intramedullary nailing with biodegradable material (BESIN) has been developed. The nails are tapped into the medullary cavity and left in place. The aim of this study was to compare BESIN technique with ESIN.

This is a prospective, randomized, controlled clinical trial including the patients (aged 5-15 years) who required operative treatment for forearm shaft fractures in two pediatric trauma centers, in Finland. The patients were randomized to be treated by BESIN or ESIN. Thirteen patients were required for each group, according to power analysis but altogether 35 were enrolled for potential drop-outs. Biodegradable polylactide-co-glycolide (PLGA) nails (ActivaNail ®, Bioretec ltd, Finland) were used in 19 and titanium nails (TEN ®, Synthes ltd, USA) in 16 patients. Pain and the range of motion (ROM) of forearm, elbow and wrist were primary outcomes. Radiographs and potential complications were analyzed of all and magnetic resonance imagines (MRI) of a randomly selected subgroup in BESIN group (N=13).

ELIGIBILITY:
Inclusion Criteria:

* suffering from single- or both-bone forearm shaft fracture
* child patient , age from 5 to 15 years
* surgical fixation needed, fracture is unstable
* cast immobilization is not rigid enough for the fracture treatment

Exclusion Criteria:

* open fractures with significant soft-tissue injury
* pathological fractures
* if patient has a previous fracture or infection in the same forearm
* patients with metabolic bone diseases, systematic disease
* patient uses the medication affecting bone quality
* resistance to infection
* fractures older than 7 days

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2011-02-20 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
The range of motion (ROM) of forearm measured by goniometer | 2 years
  The ROMs of forearm

SECONDARY OUTCOMES:
The range of motion (ROM) of elbow and wrist measured by goniometer | 2 years
  The ROMs of elbow and wrist
Pain measured with visual analogue scale | 2 years
  general pain or pain at the fracture site in mm +/- SD , scale is from 0-100mm in visual scale where child can point the proper level of pain. 0 equals "no pain", 100 equals "the highest imaginable pain"
Radiographic bone union | 2 years
  plain radiographs in anterior posterior (AP) and lateral projections
Radiographic bone deformity | 2 years
  plain radiographs in anterior posterior and lateral projections
Magnetic resonance imagining, bone healing | 2 years
  MRIs in intervention group
Implant degeneration in Magnetic resonance imagining | 2 years
  degrading of the implant
Magnetic resonance imagining, soft tissue reaction | 2 years
  soft tissue reaction

OTHER OUTCOMES:
adverse events | 2 years
  all implant or treatment related adverse events like tissue reactions or re-factures

CONTACTS AND LOCATIONS:
Overall Officials: Juhani Merikanto, Ph.D. associate professor, Principal Investigator — Central Finland, Central Hospital, Tampere, Finland
Locations (1):
- Oulu University Hospital, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baldwin K, Morrison MJ 3rd, Tomlinson LA, Ramirez R, Flynn JM. Both bone forearm fractures in children and adolescents, which fixation strategy is superior - plates or nails? A systematic review and meta-analysis of observational studies. J Orthop Trauma. 2014 Jan;28(1):e8-e14. doi: 10.1097/BOT.0b013e31829203ea. PMID 23542745
- [Background] Bostman O, Makela EA, Tormala P, Rokkanen P. Transphyseal fracture fixation using biodegradable pins. J Bone Joint Surg Br. 1989 Aug;71(4):706-7. doi: 10.1302/0301-620X.71B4.2549074. No abstract available.
- [Background] Branch LG, Crantford C, Cunningham T, Bharti G, Thompson J, Couture D, David LR. Long-Term Outcomes of Pediatric Cranial Reconstruction Using Resorbable Plating Systems for the Treatment of Craniosynostosis. J Craniofac Surg. 2017 Jan;28(1):26-29. doi: 10.1097/SCS.0000000000003166. PMID 27831975
- [Background] Garg NK, Ballal MS, Malek IA, Webster RA, Bruce CE. Use of elastic stable intramedullary nailing for treating unstable forearm fractures in children. J Trauma. 2008 Jul;65(1):109-15. doi: 10.1097/TA.0b013e3181623309. PMID 18580539
- [Background] Gorter EA, Vos DI, Sier CF, Schipper IB. Implant removal associated complications in children with limb fractures due to trauma. Eur J Trauma Emerg Surg. 2011 Dec;37(6):623-7. doi: 10.1007/s00068-011-0087-4. Epub 2011 Mar 17. PMID 22207879
- [Background] Helenius I, Lamberg TS, Kaariainen S, Impinen A, Pakarinen MP. Operative treatment of fractures in children is increasing. A population-based study from Finland. J Bone Joint Surg Am. 2009 Nov;91(11):2612-6. doi: 10.2106/JBJS.H.01519. PMID 19884435
- [Background] Herman MJ, Marshall ST. Forearm fractures in children and adolescents: a practical approach. Hand Clin. 2006 Feb;22(1):55-67. doi: 10.1016/j.hcl.2005.10.003. PMID 16504778
- [Background] Hope PG, Williamson DM, Coates CJ, Cole WG. Biodegradable pin fixation of elbow fractures in children. A randomised trial. J Bone Joint Surg Br. 1991 Nov;73(6):965-8. doi: 10.1302/0301-620X.73B6.1659570.
- [Background] Hughes TB. Bioabsorbable implants in the treatment of hand fractures: an update. Clin Orthop Relat Res. 2006 Apr;445:169-74. doi: 10.1097/01.blo.0000205884.81328.cc. PMID 16505724
- [Background] Korhonen J, Sinikumpu JJ, Harmainen S, Ryhanen J, Kallio P, Serlo W. [Removal of osteosynthesis material in children and young people]. Duodecim. 2014;130(7):689-95. Finnish. PMID 24772785
- [Background] Lascombes P, Nespola A, Poircuitte JM, Popkov D, de Gheldere A, Haumont T, Journeau P. Early complications with flexible intramedullary nailing in childhood fracture: 100 cases managed with precurved tip and shaft nails. Orthop Traumatol Surg Res. 2012 Jun;98(4):369-75. doi: 10.1016/j.otsr.2011.11.011. Epub 2012 May 14. PMID 22583892
- [Background] Lieber J, Schmittenbecher P. Developments in the treatment of pediatric long bone shaft fractures. Eur J Pediatr Surg. 2013 Dec;23(6):427-33. doi: 10.1055/s-0033-1360460. Epub 2013 Dec 10. PMID 24327219
- [Background] Makki D, Matar HE, Webb M, Wright DM, James LA, Ricketts DM. Elastic stable intramedullary nailing in paediatric forearm fractures: the rate of open reduction and complications. J Pediatr Orthop B. 2017 Sep;26(5):412-416. doi: 10.1097/BPB.0000000000000408. PMID 27832017
- [Background] Middleton JC, Tipton AJ. Synthetic biodegradable polymers as orthopedic devices. Biomaterials. 2000 Dec;21(23):2335-46. doi: 10.1016/s0142-9612(00)00101-0. PMID 11055281
- [Background] Prakasam M, Locs J, Salma-Ancane K, Loca D, Largeteau A, Berzina-Cimdina L. Biodegradable Materials and Metallic Implants-A Review. J Funct Biomater. 2017 Sep 26;8(4):44. doi: 10.3390/jfb8040044. PMID 28954399
- [Background] Sinikumpu JJ, Lautamo A, Pokka T, Serlo W. The increasing incidence of paediatric diaphyseal both-bone forearm fractures and their internal fixation during the last decade. Injury. 2012 Mar;43(3):362-6. doi: 10.1016/j.injury.2011.11.006. Epub 2011 Dec 6. PMID 22154046
- [Background] van der Eng DM, Schep NW, Schepers T. Bioabsorbable Versus Metallic Screw Fixation for Tibiofibular Syndesmotic Ruptures: A Meta-Analysis. J Foot Ankle Surg. 2015 Jul-Aug;54(4):657-62. doi: 10.1053/j.jfas.2015.03.014. Epub 2015 May 8. PMID 25960058
- [Background] Wall L, O'Donnell JC, Schoenecker PL, Keeler KA, Dobbs MB, Luhmann SJ, Gordon JE. Titanium elastic nailing radius and ulna fractures in adolescents. J Pediatr Orthop B. 2012 Sep;21(5):482-8. doi: 10.1097/BPB.0b013e3283528db5. PMID 22415404
- [Background] Waris E, Konttinen YT, Ashammakhi N, Suuronen R, Santavirta S. Bioabsorbable fixation devices in trauma and bone surgery: current clinical standing. Expert Rev Med Devices. 2004 Nov;1(2):229-40. doi: 10.1586/17434440.1.2.229. PMID 16293043
- [Result] Barber FA, Spenciner DB, Bhattacharyya S, Miller LE. Biocomposite Implants Composed of Poly(Lactide-co-Glycolide)/beta-Tricalcium Phosphate: Systematic Review of Imaging, Complication, and Performance Outcomes. Arthroscopy. 2017 Mar;33(3):683-689. doi: 10.1016/j.arthro.2016.09.032. Epub 2016 Dec 18. PMID 27998641
- [Result] Andaloussi S, Amine Oukhouya M, Alaoui O, Atarraf K, Chater L, Afifi MA. [Elastic stable intramedullary nailing (ESIN) in the treatment of both-bone forearm fractures in the child: about 87 cases]. Pan Afr Med J. 2017 May 30;27:68. doi: 10.11604/pamj.2017.27.68.11058. eCollection 2017. French. PMID 28819489
- [Result] Cullen MC, Roy DR, Giza E, Crawford AH. Complications of intramedullary fixation of pediatric forearm fractures. J Pediatr Orthop. 1998 Jan-Feb;18(1):14-21. PMID 9449095
- [Result] Dave MB, Parmar KD, Sachde BA. The Radial Bow following Square Nailing in Radius and Ulna Shaft Fractures in Adults and its Relation to Disability and Function. Malays Orthop J. 2016 Jul;10(2):11-15. doi: 10.5704/MOJ.1607.003. PMID 28435555
- [Result] Fernandez FF, Langendorfer M, Wirth T, Eberhardt O. Failures and complications in intramedullary nailing of children's forearm fractures. J Child Orthop. 2010 Apr;4(2):159-67. doi: 10.1007/s11832-010-0245-y. Epub 2010 Feb 24. PMID 21455473
- [Result] Firl M, Wunsch L. Measurement of bowing of the radius. J Bone Joint Surg Br. 2004 Sep;86(7):1047-9. doi: 10.1302/0301-620x.86b7.14294. PMID 15446536
- [Result] Krucinska I, Zywicka B, Komisarczyk A, Szymonowicz M, Kowalska S, Zaczynska E, Struszczyk M, Czarny A, Jadczyk P, Uminska-Wasiluk B, Rybak Z, Kowalczuk M. Biological Properties of Low-Toxicity PLGA and PLGA/PHB Fibrous Nanocomposite Implants for Osseous Tissue Regeneration. Part I: Evaluation of Potential Biotoxicity. Molecules. 2017 Nov 29;22(12):2092. doi: 10.3390/molecules22122092. PMID 29186078
- [Result] Kruppa C, Bunge P, Schildhauer TA, Dudda M. Low complication rate of elastic stable intramedullary nailing (ESIN) of pediatric forearm fractures: A retrospective study of 202 cases. Medicine (Baltimore). 2017 Apr;96(16):e6669. doi: 10.1097/MD.0000000000006669. PMID 28422876
- [Result] Sarmiento A, Ebramzadeh E, Brys D, Tarr R. Angular deformities and forearm function. J Orthop Res. 1992 Jan;10(1):121-33. doi: 10.1002/jor.1100100115. PMID 1727932
- [Result] Sinikumpu JJ, Keranen J, Haltia AM, Serlo W, Merikanto J. A new mini-invasive technique in treating pediatric diaphyseal forearm fractures by bioabsorbable elastic stable intramedullary nailing: a preliminary technical report. Scand J Surg. 2013;102(4):258-64. doi: 10.1177/1457496913490459. Epub 2013 Sep 20. PMID 24056134
- [Result] Sinikumpu JJ, Lautamo A, Pokka T, Serlo W. Complications and radiographic outcome of children's both-bone diaphyseal forearm fractures after invasive and non-invasive treatment. Injury. 2013 Apr;44(4):431-6. doi: 10.1016/j.injury.2012.08.032. Epub 2012 Sep 15. PMID 22986071
- [Result] Tarr RR, Garfinkel AI, Sarmiento A. The effects of angular and rotational deformities of both bones of the forearm. An in vitro study. J Bone Joint Surg Am. 1984 Jan;66(1):65-70. PMID 6690445
- [Result] Wilkins KE. Principles of fracture remodeling in children. Injury. 2005 Feb;36 Suppl 1:A3-11. doi: 10.1016/j.injury.2004.12.007. PMID 15652934
- [Result] Xue AS, Koshy JC, Weathers WM, Wolfswinkel EM, Kaufman Y, Sharabi SE, Brown RH, Hicks MJ, Hollier LH Jr. Local foreign-body reaction to commercial biodegradable implants: an in vivo animal study. Craniomaxillofac Trauma Reconstr. 2014 Mar;7(1):27-34. doi: 10.1055/s-0033-1364199. Epub 2014 Jan 9. PMID 24624254

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2018-02-05): https://cdn.clinicaltrials.gov/large-docs/00/NCT03474900/Prot_ICF_000.pdf